CLINICAL TRIAL: NCT05200598
Title: Cardiovascular Risk Predictors in Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Olga Mironova, Associate Professor, I.M. Sechenov First Moscow State Medical University
Other Study IDs: 22-21
Record Dates: First submitted 2022-01-01; First posted 2022-01-21 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Psoriasis; Cardiovascular Diseases
Keywords: psoriasis; cardiovascular risk; risk factors
MeSH Terms: conditions — Psoriasis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mild psoriasis
- Moderate psoriasis
- Severe psoriasis
- Patients without psoriasis

SUMMARY:
The investigators are planning to find the right modification of traditionally used risk scores (PASI, DLQI) in patients with psoriasis of different severity to guide the treatment that could potentially extend life, improve cardiovascular outcomes and quality of life in patients with psoriasis and cardiovascular risk factors in a prospective observational study. The traditionally excluded groups of older patients with diabetes mellitus, decreased kidney function and those with potentially worse prognosis are going to be included in the study. As it's known, the number of those patients is on the rise each year and require a close attention of multidisciplinary teams.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Written informed consent of the patient to participate in the study

Exclusion Criteria:

* Age under 18
* Pregnancy, lactation
* Very high cardiovascular risk
* Life-threatening, independently influencing prognosis and disabling diseases,
* Mental disorders that do not allow to give informed consent or answer questions adequately
* Refuse of the patient to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Considering the different severity of psoriasis, it is possible to divide patients with psoriasis into several subgroups: patients with mild psoriasis; patients with moderate psoriasis; patients with severe psoriasis who are not receiving systemic therapy; patients with severe psoriasis receiving systemic therapy with genetic-engineering biological drugs; patients with psoriatic arthritis receiving genetic-engineering biological drugs.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
SCORE2-OP risk (Systematic COronary Risk Evaluation2- Older Person) | 1 year
  Increased cardiovascular risk over the follow-up period (from low to very high)

SECONDARY OUTCOMES:
Overall mortality | 1 year
  Number of deaths due to all reasons
Cardiovascular mortality | 1 year
  Number of deaths due to cardiovascular reasons
Progression of psoriasis (PASI) | 1 year
  Progression of severity of psoriasis according to PASI (The Psoriasis Area and Severity Index - 0 to 4, none to very severe) score
Quality of life (DLQI score) | 1 year
  Impact on quality of life by DLQI (Dermatology Life Quality Index - 0 to 30, no to extremely large impact) score
Hospitalization due to cardiovascular reasons | 1 year
  Number of patients hospitalized due to cardiovascular reasons

CONTACTS AND LOCATIONS:
Overall Officials: Olga Mironova, MD, PhD, Principal Investigator — Sechenov University
Locations (1):
- University Clinical Hospital #2, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided